CLINICAL TRIAL: NCT00050076
Title: A Phase II, Double-Blind, Randomized, Exploratory, Placebo-Controlled Study of Efficacy, Safety, and Tolerability of MCC-135 Comparing QD vs BID Doses in Subjects With Congestive Heart Failure, NYHA Class II/III
Brief Title: Safety and Efficacy Study of Once and Twice Daily Doses of MCC-135 in Subjects With Congestive Heart Failure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-02-TL-MCC135-001; U1111-1127-6077 (Registry Identifier: WHO)
Record Dates: First submitted 2002-11-20; First posted 2002-11-21 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Cardiac Failure; Heart Decompensation; Drug Therapy
MeSH Terms: conditions — Heart Failure | interventions — MCC 135

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MCC-135 50 mg BID (Experimental)
  Interventions: Drug: MCC-135
- MCC-135 100 mg QD (Experimental)
  Interventions: Drug: MCC-135
- MCC-135 200 mg QD (Experimental)
  Interventions: Drug: MCC-135
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCC-135 — MCC-135 50 mg, tablets, orally, twice daily for up to 12 weeks
  Arms: MCC-135 50 mg BID
Drug: MCC-135 — MCC-135 100 mg, tablets, orally, once daily for up to 12 weeks
  Arms: MCC-135 100 mg QD
Drug: MCC-135 — MCC-135 200 mg, tablets, orally, once daily for up to 12 weeks
  Arms: MCC-135 200 mg QD
Drug: Placebo — MCC-135 placebo-matching tablets, orally, once daily for up to 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of two different doses of MCC-135, once daily (QD) or twice daily (BID), on the disease state and the quality of life in subjects with congestive heart failure.

DETAILED DESCRIPTION:
In recent years the usefulness of angiotensin converting enzyme inhibitors and vasodilators as well as beta-blockers has been realized in the treatment of heart failure. Multi-center studies clinical trials have shown some benefit of angiotensin converting enzyme inhibitors on the morbidity and mortality of heart failure subjects, and physicians are also prescribing angiotensin converting enzyme inhibitors for the initial treatment of subjects with left ventricular dysfunction. Some subjects do not respond to angiotensin converting enzyme inhibitors and intolerance to these compounds has also been observed. Despite the significant reduction in mortality observed in limited controlled studies, the 5-year mortality of subjects with congestive heart failure continues to be high, indicating that there is a significant therapeutic gap in the treatment of this disease.

MCC-135 is being studied to assess its usefulness as a supplement or replacement to current treatment and to provide subjects with specific and predictable therapy that will reverse the remodeling of the diseased heart and markedly improve the subject's survival. The current study is an exploratory clinical trial to determine the efficacy of two doses and two dose regimens of MCC-135 when compared to placebo by evaluating improvement in the subject's plasma b-type (brain) natriuretic peptide levels, regular rate (heart rate) variability and clinical signs and symptoms.

ELIGIBILITY:
Inclusion:

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Having a clinical diagnosis consistent with congestive heart failure, of at least 6 months duration and clinically stable for the last month.
* Has a left ventricular ejection fraction less than or equal to 40%.
* Has Plasma b-type (brain) natriuretic peptide levels greater than or equal to 200 pg/ml at screening.
* Meeting the following requirements for current concomitant medication:

  * Must be using an angiotensin converting enzyme inhibitor or Angiotensin II receptor antagonists therapy for at least 1 month prior to the screening visit.
  * If using beta-blockers, must have commenced treatment at least 4 months prior to the screening visit.
  * All other cardiac medications must have been introduced at least one month prior to the screening visit.

Exclusion:

* Heart failure primarily due to:

  * Obstructive valvular disease
  * Malfunctioning artificial heart valve
  * Congenital heart disease
  * Pericardial disease
  * Uncontrolled thyroid disease
  * Amyloidosis
  * Severe pulmonary disease
  * Restrictive or obstructive cardiomyopathy
  * Known active myocarditis
* Terminal heart failure or on waiting list for transplant.
* Atrio-ventricular block except for first-degree atrio-ventricular block.
* A history of or currently sustained ventricular tachycardia.
* Subjects with atrial fibrillation and/or requiring pacemakers (including bi-ventricular pacing).
* Presence of pulmonary embolism.
* Acute myocardial infarction, unstable angina, coronary revascularization or major surgery during the last 6 weeks prior to screening.
* Episode of syncope or cardiac arrest during the last 6 weeks prior to screening.
* Requiring treatment with the following therapies:

  * Anti-arrhythmics (Amiodarone/beta-blockers are permitted)
  * Calcium sensitizers
  * Catecholamines
  * Phosphodiesterase inhibitors
* Is currently participating in another investigational study or who have participated in an investigational study (including MCC-135) during the 2 months prior to the screening visit
* Has a history of drug or alcohol abuse, as defined by Diagnostic and Statistical Manual of Mental Disorders-4th edition criteria, within the past two years.
* Has significant, moderate-severe renal dysfunction or disease, confirmed by serum creatinine of greater than 2mg/dl (180 micromol/L).
* Serum potassium levels at entry confirmed below 3.5mmol/L.
* Known severe symptomatic primary pulmonary disease in the last 5 years e.g. asthma, chronic obstructive pulmonary disease.
* Concurrent severe disease (including significant hepatic, metabolic or other systemic disease) or any medical condition that, in the opinion of the investigator, would compromise the subject's safety or their successful participation in the study.
* History of multiple drug allergies or with a known allergy to the study drug or any medicine chemically related to the study drug.
* Individuals who are morbidly obese.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Anti-arrhythmics (Amiodarone/beta-blockers are permitted)
  * Calcium sensitizers
  * Catecholamines
  * Phosphodiesterase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2002-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the serum levels of brain natriuretic peptide | At Final Visit.

SECONDARY OUTCOMES:
Change from baseline in the Minnesota living with heart failure questionnaire score | At Final Visit.
Regular rate (heart rate) variability as measured by 24-hour Holter monitoring | At Final Visit.
Disease progression status measured by New York Heart Association class | At Final Visit.
Disease progression status measured by Global Clinical Status | At Final Visit.
Disease progression status measured by Clinical Composite | At Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (53):
- United States (53):
  - Maricopa Medical Center, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Capitol Intervention Cardiology, Carmichael, California
  - San Diego Cardiovascular, Encinitas, California
  - LAC & USC Medical Center, Los Angeles, California
  - ARI Clinical Trials, Inc Arrhythmia Research & Cardiology Health Center, Redondo Beach, California
  - Clinical Trials Research, Roseville, California
  - Sacramento Heart & Vascular Medical Associates, Sacramento, California
  - University of California San Diego, San Diego, California
  - Apex Research Institute, Santa Ana, California
  - Cardiology Consultants PA, Daytona Beach, Florida
  - Cardiology Associates of Fort Lauderdale, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Southern Clinical Research & Management, Augusta, Georgia
  - Medical Group of Fort Wayne, PC, Fort Wayne, Indiana
  - Medical Center Cardiologist, Louisville, Kentucky
  - Louisville Cardiology Medical Group, PSC, Louisville, Kentucky
  - Louisiana Heart Center, Chalmette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Cardiac Center of Louisiana, LLC, Shreveport, Louisiana
  - Cardiology Associates, PC, Annapolis, Maryland
  - University of Maryland Hospital, Baltimore, Maryland
  - Cardiovascular Consultants, PA, Takoma Park, Maryland
  - University of Massachusettes, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Millburn, New Jersey
  - South Jersey Heart Group, Sewell, New Jersey
  - Buffalo General Hospital, Buffalo, New York
  - Heart Care Center East, Fayetteville, New York
  - Hudson Valley Clinical Research, Kingston, New York
  - Saint Vincent Catholic Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Sterling Research Group, Cincinnati, Ohio
  - North Ohio Research, Ltd., Lorain, Ohio
  - City Cardiology Associates, Inc., Stow, Ohio
  - Chestnut Hill Cardiology, Ltd., Flourtown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Research Associates, Columbia, South Carolina
  - The Stern Cardiovascular Center, Memphis, Tennessee
  - Cardiovascular Research Institute of Dallas Medical Center - Cardiologist Research Foundation, Dallas, Texas
  - Med-Tech Research, Houston, Texas
  - Nassau Bay, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Cardiovascular Associates, Ltd., Chesapeake, Virginia
  - Wisconsin Center for Clinical Research, LLC, Elkhorn, Wisconsin